CLINICAL TRIAL: NCT01808482
Title: A First Time in Human Study Exploring Preliminary Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK2618960 in Healthy Volunteers and Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: A First Time in Human Study Exploring Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of GSK2618960 in Healthy Volunteers and Patients With Relapsing Remitting Multiple Sclerosis (RRMS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: GSK confirmed misrepresentation of preclinical data that supported the rationale for GSK2618960 in MS. This decreased benefit assessment for MS
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 116702
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: monoclonal antibody; Multiple Sclerosis; Interleukin-7 Receptor
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — GSK2618960

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part A: GSK2618960 (Experimental): Subjects will receive ascending single dose in 3:1 ratio of active:placebo respectively in each dosing session.
  Interventions: Drug: Part A: 100 mg/mL GSK2618960
- Part A: Placebo (Placebo Comparator): Subjects will receive ascending single dose in 3:1 ratio of active:placebo respectively in each dosing session
  Interventions: Drug: Part A: matching placebo
- Part B: GSK2618960 (Experimental): Subjects will receive ascending repeat dose (dose decided from Part A) in 3:1 ratio of active:placebo respectively in each cohort.
  Interventions: Drug: Part B: Dose of GSK2618960 decided from Part A
- Part B: Placebo (Placebo Comparator): Subjects will receive ascending repeat dose (dose decided from Part A) in 3:1 ratio of active:placebo respectively in each cohort.
  Interventions: Drug: Part B: matching placebo
- Part C: GSK2618960 (Experimental): Subjects will receive active treatments for 2 to 4 repeated doses (dose decided from Part A& B)
  Interventions: Drug: Part C: Dose of GSK2618960 decided from Part A and B

INTERVENTIONS:
Drug: Part A: 100 mg/mL GSK2618960 — 100 mg/mL GSK2618960 solution for IV Infusion up to 1 hr except for the 1st dose (IV bolus) and 2nd dose (IV infusion over 5 min) of Part A
  Arms: Part A: GSK2618960
Drug: Part A: matching placebo — Matching placebo
  Arms: Part A: Placebo
Drug: Part B: Dose of GSK2618960 decided from Part A — 100 mg/mL GSK2618960 solution for IV Infusion in repeat dose decided from Part A
  Arms: Part B: GSK2618960
Drug: Part B: matching placebo — Matching placebo
  Arms: Part B: Placebo
Drug: Part C: Dose of GSK2618960 decided from Part A and B — 100 mg/mL GSK2618960 solution for IV Infusion in repeat dose decided from Part A and B
  Arms: Part C: GSK2618960

SUMMARY:
This is a 3-part study where Parts A, B (single-blind - investigator and subject blind) will enrol healthy volunteers and Part C (open-label) will enrol RRMS patients. Parts A (single ascending dose) and B (repeat ascending dose) will assess safety, tolerability, PK and PD of GSK2618960. Part C (repeat doses) will assess safety, tolerability, PK, PD, immunogenicity, paraclinical (magnetic resonance imaging [MRI] lesion counts) disease activity and markers of Th1 and Th17 mechanisms.

Part A: Each of the 24 healthy volunteers (divided in 5 groups), will take part in only 2 of the planned 8 dosing sessions (A-active, P-placebo). Subjects in each group of Part A will be randomized in a 2:1:1 ratio to one of the following sequences: AA, AP or PA such that in each dosing session they will receive study treatment in a 3:1 ratio of active: placebo respectively.

Part B: Dosing levels and regimen are dependent upon safety tolerability and PK/receptor occupancy (RO) data from Part A. In Cohort 1, 12 subjects will be randomized in a 3:1 ratio to A or P. Each subject will receive the same study treatment for repeated doses. If the duration of full RO from highest dose in Part A is less than 4 weeks, a second cohort of 12 subjects in Part B may be recruited, based on Dose Escalation Committee (DEC) decision Part C: The 20 RRMS patients will be assigned to active treatments for 2 to 4 repeated doses.

Safety/tolerability and PK data monitoring and the decision to proceed to the next dose level of GSK2618960, and the decisions to proceed to Part B and Part C of the study will be made by a dose escalation committee.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

* Healthy as determined by a responsible and experienced physician
* Male between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Alanine aminotransferase (ALT), alkaline phosphatase (AP) and bilirubin <=1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Corrected QT interval using Fridericia's (QTcF) < 450 milliseconds (msec).
* Body weight >=50 kilogram (kg), <=100 kg and body mass index (BMI) within the range 19.0 - 29.9 kg/meter squared (m^2) (inclusive).
* Subjects with history of current vaccination status for tetanus, diphtheria, pertussis, measles, mumps and rubella (or consent to vaccination at screening). Subjects with history of current vaccination status for influenza or who consent to receive influenza vaccine at screening if study dosing is predicted to result in >75% RO during Flu season (October - April).
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study.

MS Patients

* Suitable as determined by the Principal Investigator, based on his/her overall evaluation.
* Must have a confirmed diagnosis of RRMS according to 2010 revisions to McDonald Criteria..
* Must have a history of at least two clinical episodes of demyelination.
* Have demonstrated clinical or paraclinical activity in 12 months prior to screening (which may have occurred whilst on a disease-modifying therapy) by either: One or more documented relapses,OR one or more documented Gd enhancing lesions in the brain or spinal cord,
* Expanded Disability Status Scale (EDSS) score <=0 at the screening.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate as follows: Non-childbearing potential, females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods and women of childbearing potential should have used one of the contraception methods.
* Male subjects must agree to use one of the contraception methods.
* Subjects with history of current vaccination status for tetanus, diphtheria, pertussis, measles, mumps and rubella (or who consent to vaccination at screening). Subjects with expected study participation during Flu season (October - April) only, with history of current vaccination status for influenza or consent to receive influenza vaccine at screening.
* Body weight >=50 kg.
* On ECG, QTcF interval <450 msec; or QTcF <480 msec in subjects with bundle branch block.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form, and authorisation of the release and use of protected health information (PHI).

Exclusion Criteria:

Healthy Volunteers

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* History of smoking within 6 months of screening.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males. One unit is equivalent to 8 g of alcohol: a half-pint (~240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other significant allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Subjects, who in the investigator's judgement, pose a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behaviour in the last 6 months and/or any suicidal ideation of type 4 or 5 on the C-SSRS in the last 2 months.
* Previous history of anaphylaxis and severe allergic reaction.
* Receipt of live vaccination within 1 month of screening (excluding flu vaccination) or plan to receive live vaccination during the study.

MS Patients

* Intolerant, or unwilling, to undergo MRI scanning.
* Contraindications for administration of Gd-contrast agents i.e. history of allergy to gadolinium.
* Subjects, who in the investigator's judgement, pose a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behaviour in the last 6 months and/or any suicidal ideation of type 4 or 5 on the C-SSRS in the last 2 months.
* History of, or laboratory findings indicative of any clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic (other than MS), dermatologic, psychiatric, renal, and/or other major disease or of known drug sensitivity that would preclude the administration of a recombinant humanized antibody or the use of systemic steroids during the course of the study.
* Abnormal baseline blood tests exceeding any of the limits defined below: ALT or aspartate transaminase (AST) >1.5 x the ULN, AP and bilirubin >1.5X ULN (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%), total white blood cell count <2,500/millimetre cube (mm^3), if lymphocyte count is less than the Lower Limit of Normal (LLN), maybe included only if PI and GSK Medical Monitor agree that doesn't introduce additional risk, platelet count < 95,000/mm3, creatinine >2 x ULN, calculated creatinine clearance <60 ml/min (per Cockcroft & Gault) at Screening, International Normalised Ratio (INR) larger than upper limit of the normal reference range (0.9 - 1.3).

A subject with a clinical abnormality or laboratory parameters significantly outside the above reference range for the population being studied may be included only if the Investigator and the GlaxoSmithKline Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.

* Treatment with methylprednisolone or any other systemic steroid, for a relapse or otherwise, within 30 days of dosing.
* Treatment with first line disease modifying therapies for RRMS, such as glatiramer acetate or beta-interferons within 6 weeks prior to screening.
* Treatment within the past 12 months or currently with any of the following agents: cyclosporine, cladribine, natalizumab (Tysabri) or other monoclonal antibodies, murine protein, T-cell vaccination, plasmapheresis, intravenous (IV) Immunoglobulin G (IgG), stem cell transplantation.
* Treatment in the past 6 months with any of the following agents: Fingolimod (Gilenya), methotrexate, mitoxantrone, azathioprine, or other small molecule immunosuppressants.
* History of intolerance to paracetamol, ibuprofen, naproxen or other non-steroidal anti-inflammatory agents which would preclude use of at least one of these during the study.
* Previous history of anaphylaxis, severe allergic reaction, generation of neutralizing antibodies, or hypersensitivity to albumin or a protein-based therapeutic, including natalizumab (Tysabri) or any other monoclonal antibody.
* A positive pre-study hepatitis B surface antigen or positive hepatitis C antibody result.
* Known diagnosis or history consistent with human immunodeficiency virus (HIV) positivity
* Subjects with evidence of dementia or psychiatric illness which, in the Investigator's opinion, is likely to prevent them from a full understanding of and/or compliance with the study requirements and procedures. .
* Blood donation (1 unit or more) within 3 months prior to investigational drug administration.
* History of regular alcohol consumption within 6 months of the study defined as:

Average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.

* Subjects who have received live vaccinations 1 month prior to screening (excluding flu vaccination) or plan to receive live vaccination during the study.
* Smokers unable to abstain from smoking while on the clinical unit.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2013-08-06 (Actual); Study Completion 2013-08-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSK2618960 as assessed by changes in: vital signs, ECG monitoring, haematology, clinical chemistry, urinalysis, and monitoring of AEs in healthy volunteers and MS patients | Upto Week 12 pending emerging data and DEC decisions.
  Safety and tolerability parameters will include recording of vital signs, electrocardiogram (ECG)s, safety labs, and adverse event (AE)s, in Part A/B/C of the study in healthy volunteers and Multiple Sclerosis (MS) patients.
Safety and tolerability of GSK2618960 as assessed by changes in MS relapses: Number, duration, severity in MS patients | Upto Week 12 pending emerging data and DEC decisions
  Safety and tolerability parameters will include recording of the number/duration/severity of MS relapses in Part C of the study in MS patients

SECONDARY OUTCOMES:
Composite of PK parameters of GSK2618960 | Day 1 predose 1,2,4, 8, 24 hour (hr)s post dose (Day 2), 36 hrs (Day 2), Day 3, Day 4, Day 8, Day 15, and post Day 15 every 2 weeks and dependent upon predictions.
  The following pharmacokinetic (PK) data will be calculated: maximum concentration (Cmax), area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration [AUC(0-tau)] and AUC from zero to infinity [AUC(0-inf)], percentage of AUC(0-inf) obtained by extrapolation (%AUC(ex)), clearance (CL), volume of distribution (Vss), time from administration to Cmax (tmax) and elimination half life (t½) of GSK2618960.
Receptor occupancy by GSK2618960 - Blinding of fluorophore-conjugated competing and non-competing antibody of GSK2618960 following the single and repeat IV doses | Day 1 predose 1, 4, 8 hrs dose, Day 2, Day 3, Day 4, Day 8, Day 15, and Day 29 onwards visits through final follow up, and dependent upon predictions.
  The total receptor levels will be measured by counting the binding of fluorophore-conjugated competing antibody (PE-GSK2618960) to unoccupied GSK2618960 binding sites, normalized by baseline and maximum blocking controls, in addition to non-competing antibody binding.
Relationship between dose and duration of >95% RO of GSK2618960 following single and repeat IV doses in healthy volunteers | Day 1 predose 1,2,4, 8, 24 hour (hr)s post dose (Day 2), 36 hrs (Day 2), Day 3, Day 4, Day 8, Day 15, and post Day 15 every 2 weeks and dependent upon predictions.
  The PK/RO relationship of GSK2618960 following single and repeat IV doses in Part A and B of the study.
To characterize the effect of GSK2618960 on IL-7 downstream signalling - Phosphorylation level of stat5 protein upon ex vivo stimulation of IL-7 cytokine, normalized by baseline, maximum receptor blocking controls and unstimulated controls | Day -1, Day 8, Day 15 and Day 29 onwards through final follow up, dependent upon predictions.
  Blood from 7 distinct healthy donors was incubated ex vivo with 0.003 to 100 microgram/mL GSK2618960 and then stimulated with 5ng/mL human IL-7 STAT5 phosphorylation as well as unbound GSK2618960 and total IL-7R levels were assayed by flow cytometry.
Presence of antibodies to GSK2618960 | Immunogenicity sampling will be performed at Day1 pre-dose, Day 15 and approximately 2 months after dosing for dosing sessions 1- 5, and performed every 3 months after final dosing for dosing sessions 6-8 and parts B & C.
  Presence of antibodies to GSK2618960 will be assessed in serum samples using validated ECL assays.
Changes in numbers and relevant ratios of lymphocyte subsets | Day -1, Day 8, Day 15 and Day 29 onwards through final follow up, will be dependent upon predictions.
  Lymphocyte subsets will include B cells, CD3+ T cells, NK cells, regulatory T cells, and recent thymic emigrants, and may include, CD4+T cell, CD8+ T cells, naïve CD4+ T cells, effect memory CD4+ T cells, and central memory CD4+ T cell, etc. For Part A, blood sampling for lymphocyte subset is not required for dosing sessions 1-3. For part A, after day 29, a maximum of 3 blood samples will be drawn, each separated by 2 weeks, at time points spanning the predicted end of full RO. For parts B and C, blood sampling is limited to Day -1, and 3 blood samples separated by 2 weeks.
Markers of serum inflammatory mediators in blood. | Day 1 predose and 1 h and 4 h post dose, Day 2 and Day 3
  Serum inflammatory mediators, including some or all, but not limited to: IL-1β, IL-6, IL-8, MCP-1, TNF-α and IFN-γ blood sampling for serum inflammatory mediators will be performed for dose sessions 1, 2, 3, 6; optional for other dose sessions in part A, Part B and Part C pending emerging data
Cumulative number of new brain lesions | 1st MRI baseline at -8weeks, 2nd MRI baseline at -4 weeks, 3rd MRI baseline on Day -1, and at Week 6, Week 10, Week 14 and Week 18 after first dose
  Cumulative number of new brain lesions will be assessed in Part C of the study using magnetic resonance imaging (MRI). New lesion is defined as enhancing in the presence of Gadolinium contrast agent.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 116702 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116702?search=study&study_ids=116702#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 116702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register